CLINICAL TRIAL: NCT02346201
Title: Apathy in Dementia Methylphenidate Trial 2
Acronym: ADMET2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ADMET2; R01AG046543 (NIH)
Record Dates: First submitted 2015-01-20; First posted 2015-01-26 (Estimated); Results first posted 2023-06-13 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Apathy; Alzheimer's Disease
MeSH Terms: conditions — Lethargy; Alzheimer Disease | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Methylphenidate (Active Comparator): Methylphenidate, target dose 20 mg per day (range 10-20 mg per day), in 5 mg over-capsulated tablets, and psychosocial intervention
  Interventions: Drug: Methylphenidate
- Placebo (Placebo Comparator): Matching over-encapsulated placebo and psychosocial intervention
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Methylphenidate — Two 5mg methylphenidate over-encapsulated drug taken twice a day for 6 months (total of 20 mg methylphenidate per day), and psychosocial intervention
  Other Names: Ritalin
  Arms: Methylphenidate
Drug: Placebo — Two over-encapsulated placebo taken twice a day for 6 months and psychosocial intervention
  Arms: Placebo

SUMMARY:
Apathy in Dementia Methylphenidate Trial 2 (ADMET 2) is a Phase III, placebo-controlled, masked, 6 month, multi-center randomized clinical trial sponsored by National Institutes of Aging involving 200 participants with Alzheimer's disease (AD). ADMET 2 is designed to examine the efficacy and safety of methylphenidate as treatment for clinically significant apathy in AD participants. ADMET 2 will enroll participants from real world settings such as outpatient, nursing home, and assisted living facilities and will examine the effects of methylphenidate on apathy and cognition. ADMET 2 will also conduct careful safety monitoring.

DETAILED DESCRIPTION:
ADMET 2 will examine in a masked, randomized trial the efficacy of methylphenidate for the treatment of clinically significant apathy in participants with Alzheimer's dementia. Efficacy will be assessed as the change in Neuropsychiatric Inventory Apathy subscale (NPI apathy) from baseline to 6 months and score on the Alzheimer's Disease Cooperative Study - Clinical Global Impression of Change (CGIC) scale at 6 months.

ADMET 2 will also examine the safety of methylphenidate for the treatment of clinically significant apathy in participants with Alzheimer's disease by measuring vital signs, electrolyte panels, adverse event reports, and electrocardiograms. Safety will also be measured by examining neuropsychiatric symptoms other than apathy using the Neuropsychiatric Inventory (NPI).

Changes from baseline to 6 months in other neuropsychological assessments as measured using the Dementia Apathy Interview and Rating (DAIR) scale will also be assessed.

Cost-effectiveness will be measured by assessing quality of life and economic assessment and cognitive changes using a cognitive battery that includes the Mini Mental State Exam (MMSE) and other scales.

A biomarker sub-study initiated part-way through the main trial will collect information on blood-based biomarkers, including microRNA, markers of oxidative stress, inflammation, neuronal loss and lipidomics.

ELIGIBILITY:
Inclusion criteria

* Possible or probable Alzheimer's disease (National Institute of Neurological and Communicative Disorders and Stroke - Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) criteria), with Mini-Mental State Exam (MMSE) score of 10-28 inclusive
* Clinically significant apathy for at least four weeks for which either

  * the frequency of apathy as assessed by the Neuropsychiatric Inventory (NPI) is 'Very frequently', or
  * the frequency of apathy as assessed by the NPI is 'Frequently' or 'Often' AND the severity of apathy as assessed by the NPI is 'Moderate' or 'Marked'
* A medication for apathy is appropriate, in the opinion of the study physician
* Provision of informed consent for participation in the study by potential participant or surrogate (with participant assent if the potential participant is unable to provide informed consent) and caregiver
* Availability of primary caregiver, who spends greater than ten hours a week with the potential participant and supervises his/her care, to accompany the potential participant to study visits and to participate in the study
* Sufficient fluency, of both the potential participant and caregiver, in written and spoken English to participate in study visits, physical exams, and outcome assessments
* If female, woman must be post-menopausal for at least 2 years or have had a hysterectomy

Exclusion criteria

* Currently meets criteria for Major Depressive Episode, by Diagnostic Statistical Manual of Mental Disorder - IV (TR) criteria
* Clinically significant agitation /aggression for which either

  * the frequency of agitation /aggression as assessed by the NPI is 'Very frequently', or
  * the frequency of agitation /aggression as assessed by the NPI is 'Frequently' AND the severity of the agitation as assessed by the NPI is 'Moderate', or 'Marked'
* Clinically significant delusions for which either

  * the frequency of delusions as assessed by the NPI is 'Very frequently', or
  * the frequency of delusions as assessed by the NPI is 'Frequently' AND the severity of the delusions as assessed by the NPI is 'Moderate', or 'Marked'
* Clinically significant hallucinations for which either

  * the frequency of hallucinations as assessed by the NPI is 'Very frequently', or
  * the frequency of hallucinations as assessed by the NPI is 'Frequently' AND the severity of the hallucinations as assessed by the NPI is 'Moderate', or 'Marked'
* Change to AD medications within the month preceding randomization, including starting, stopping, or dosage modifications
* Change in anti-depressant (except for trazodone used for sleeping difficulties as described below) use within the 30 days preceding randomization or a period of time equal to 5 half-lives of drug, whichever period of time is longer
* Use of trazodone > 50mg or lorazepam > 0.5mg or for indications other than sleeping difficulties within the 30 days preceding randomization or a period of time equal to 5 half-lives of drug, whichever period of time is longer. Other benzodiazepines are prohibited in the past 30 days or within 5 half-lives, whichever period of time is longer.
* Failure of treatment with methylphenidate in the past for apathy after convincing evidence of an adequate trial as judged by study physician
* Currently taking any amphetamine product, an antipsychotic, bupropion, or any medication that would prohibit the safe concurrent use of methylphenidate, including but not limited to monoamine oxidase inhibitors and tricyclic antidepressants within the 30 days preceding randomization or a period of time equal to 5 half-lives of drug, whichever period of time is longer
* Need for acute psychiatric hospitalization or is suicidal in the opinion of the study physician
* Significant communicative impairments that would affect participation in clinical trial
* Central nervous system abnormalities (e.g., cerebral aneurysm), seizures (convulsions, epilepsy), Tourette's syndrome or presence of motor tics, or abnormal electroencephalograms
* Lack of appetite that results in significant unintentional weight loss as determined by the study physician in the last three months
* Uncontrolled hyperthyroidism
* Any cardiovascular or cerebrovascular abnormality deemed to be clinically significant by the study physician, tachycardia (heart rate > 100 beats per minute), or uncontrolled hypertension (defined as medication non-compliance or past 3 months with a diastolic reading > 105 mm Hg), at the time of screening
* Closed angle glaucoma or pheochromocytoma
* Women with childbearing potential
* Current participation in a clinical trial or study that may add significant burden or affect study outcomes
* Any condition that, in the opinion of the study physician, makes it medically inappropriate or risky for the potential participant to enroll in the trial, including, but not limited to, contraindication to treatment with methylphenidate.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2016-01; Primary Completion 2020-07-15 (Actual); Study Completion 2020-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacobo Mintzer, MD, Study Chair — Medical University of South Carolina
Locations (10):
- United States (9):
  - Banner Alzheimer's Institute, Phoenix, Arizona
  - University of Arkansas, Little Rock, Arkansas
  - Yale Alzheimer's Disease Research Unit, New Haven, Connecticut
  - Emory, Atlanta, Georgia
  - Johns Hopkins University, Baltimore, Maryland
  - University of Rochester, Rochester, New York
  - Wake Forest, Winston-Salem, North Carolina
  - University Hospitals- Case Medical Center, Cleveland, Ohio
  - Roper-St. Francis Healthcare, Charleston, South Carolina
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Sankhe K, Ruthirakuhan M, Andreazza AC, Brawman-Mintzer O, Craft S, Herrmann N, Ismail Z, Lerner AJ, Levey AI, Mintzer J, Padala PR, Perin J, Porsteinsson AP, Rosenberg PB, Shade D, Tumati S, van Dyck CH, Lanctot KL. Peripheral biomarkers associated with apathy and predicting response to methylphenidate: Secondary analysis of the Apathy in Dementia Methylphenidate Trial 2 (ADMET2) study. Int Psychogeriatr. 2026 Jan 10:100181. doi: 10.1016/j.inpsyc.2025.100181. Online ahead of print. PMID 41521126
- [Derived] Lanctot KL, Chen C, Mah E, Kiss A, Li A, Shade D, Scherer RW, Vieira D, Coulibaly H, Rosenberg PB, Lerner AJ, Padala PR, Brawman-Mintzer O, van Dyck CH, Porsteinsson AP, Craft S, Levey A, Burke WJ, Mintzer J, Herrmann N. Cost consequence analysis of Apathy in Dementia Methylphenidate Trial 2 (ADMET 2). Int Psychogeriatr. 2023 Nov;35(11):664-672. doi: 10.1017/S1041610223000327. Epub 2023 Apr 17. PMID 37066690
- [Derived] Mintzer J, Lanctot KL, Scherer RW, Rosenberg PB, Herrmann N, van Dyck CH, Padala PR, Brawman-Mintzer O, Porsteinsson AP, Lerner AJ, Craft S, Levey AI, Burke W, Perin J, Shade D; ADMET 2 Research Group. Effect of Methylphenidate on Apathy in Patients With Alzheimer Disease: The ADMET 2 Randomized Clinical Trial. JAMA Neurol. 2021 Nov 1;78(11):1324-1332. doi: 10.1001/jamaneurol.2021.3356. PMID 34570180
- [Derived] Scherer RW, Drye L, Mintzer J, Lanctot K, Rosenberg P, Herrmann N, Padala P, Brawman-Mintzer O, Burke W, Craft S, Lerner AJ, Levey A, Porsteinsson A, van Dyck CH; ADMET 2 Research Group. The Apathy in Dementia Methylphenidate Trial 2 (ADMET 2): study protocol for a randomized controlled trial. Trials. 2018 Jan 18;19(1):46. doi: 10.1186/s13063-017-2406-5. PMID 29347996

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Methylphenidate | Placebo
Started | 99 | 101
Completed | 89 | 92
Not Completed | 10 | 9
Not completed — Adverse Event | 3 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 6 | 3
Not completed — Unavailable for future follow-up | 0 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Missed final visit | 0 | 2

BASELINE CHARACTERISTICS:
Population: baseline data are missing for one participant in the methylphenidate group
Groups:
- Total: Total of all reporting groups
Arm/Group | Methylphenidate | Placebo | Total
Number analyzed (Participants) | 98 | 101 | 199
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 77 [71 to 81] | 76 [70 to 81] | 76 [71 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 35 | 68
  Male | 65 | 66 | 131
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 98 | 100 | 198
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 90 | 91 | 181
  Race: Black or African American | 6 | 6 | 12
  Race: American Indian or Alaskan Native | 0 | 0 | 0
  Race: Asian | 0 | 0 | 0
  Race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Race: Other | 1 | 4 | 5
  Race: More than one race | 0 | 0 | 0
  Race: Unknown or not reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Neuropsychiatric Inventory (NPI)
Description: Mean difference in change from baseline to 6 months in the NPI apathy subscale scores as administered by certified personnel to the study caregiver.
  SEVERITY is graded 1 to 3 and FREQUENCY is graded 1 to 4. The overall score for the domain is the product of the severity and frequency which ranges from 1 to 12 with higher scores indicating more apathy.
Time Frame: baseline to 6 months
Population: The number of participants with data at 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Methylphenidate | Placebo
Number analyzed (Participants) | 89 | 91
score on a scale | -4.5 (4.1) | -3.1 (3.6)

2. Primary Outcome: Percentage of Participants With Change in Modified Alzheimer's Disease Cooperative Study- Clinical Global Impression of Change (CGIC)
Description: Percentage of individuals improving on Alzheimer's Disease Cooperative Study- Clinical Global Impression of Change (CGIC) from baseline to 6 months; the CGIC is a 7-point Likert scale used to rate each patient with the following scores: "marked worsening"(7), "moderate worsening" (6), "minimal worsening"(5), "no change"(4), "minimal improvement"(3), "moderate improvement"(2), "marked improvement"(1). Ratings were based on an interview with the caregiver and an examination of the patient. The CGIC requires the clinician to consider a number of aspects of apathy, such as level of initiative, level of interest, and emotional engagement. Reported data is the percentage of participants with minimal/moderate/marked improvement.
Time Frame: Baseline to month 6
Population: The number of participants with data at 6 months
Measure: Number; unit: percentage of participants
Arm/Group | Methylphenidate | Placebo
Number analyzed (Participants) | 89 | 91
percentage of participants | 39 | 32

ADVERSE EVENTS:
Time Frame: 6 months (enrollment until study completion)
Arm/Group | Methylphenidate | Placebo
All-Cause Mortality (participants affected / at risk) | 0/99 | 0/101
Serious Adverse Events (participants affected / at risk) | 13/99 | 9/101
Other Adverse Events (participants affected / at risk) | 97/99 | 99/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Methylphenidate (N=99) | Placebo (N=101)
Hospitalization/ER visit for confusion/weakness (Psychiatric disorders) | 3 (3) | 1 (1)
Hospitalization/ER visit for planned surgery (Surgical and medical procedures) | 3 (3) | 0 (0)
Hospitalization/ER visit for UTI/other infection (Infections and infestations) | 1 (1) | 3 (3)
Hospitalization/ER visit for Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Hospitalization/ER visit for congestive heart failure or exacerbation (Cardiac disorders) | 1 (1) | 1 (2)
Hospitalization/ER visit for weakness/fever (General disorders) | 1 (1) | 0 (0)
Hospitalization/ER visit for atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Hospitalization/ER visit for upper arm and chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hospitalization/ER visit for Bradycardia/nausea (Cardiac disorders) | 1 (1) | 0 (0)
Hospitalization/ER visit for peripheral blood clots (Vascular disorders) | 0 (0) | 1 (1)
Hospitalization/ER visit for facial drooping (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hospitalization/ER visit for multiple seizures (Nervous system disorders) | 0 (0) | 1 (1)
Hospitalization/ER visit for abdominal pain and constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hospitalization/ER visit for cholecystitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hospitalization/ER visit for diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hospitalization/ER visit for gait impairment and transient visual loss (General disorders) | 1 (1) | 0 (0)
Hospitalization/ER visit for syncope (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Methylphenidate (N=99) | Placebo (N=101)
Abdominal pain (Gastrointestinal disorders) | 17 | 12
aggressive behavior or hostility (Psychiatric disorders) | 26 | 27
Agitation (Nervous system disorders) | 45 | 53
Anemia (Blood and lymphatic system disorders) | 7 | 3
angina (Cardiac disorders) | 5 | 5
anorexia (Metabolism and nutrition disorders) | 20 | 16
anxiety, nervousness, or tension (Nervous system disorders) | 41 | 52
arthralgia (Musculoskeletal and connective tissue disorders) | 40 | 42
blood pressure changes (Vascular disorders) | 15 | 9
blurry vision or eyesight changes (Eye disorders) | 14 | 14
decreased appetite (Metabolism and nutrition disorders) | 32 | 31
depressed mood (Psychiatric disorders) | 35 | 40
distractibility (Social circumstances) | 42 | 35
dizziness (Ear and labyrinth disorders) | 24 | 20
drowsiness (General disorders) | 43 | 44
dry mouth (Gastrointestinal disorders) | 22 | 19
dyskinesia (Nervous system disorders) | 10 | 8
fever (General disorders) | 7 | 5
hair loss (Endocrine disorders) | 6 | 7
headache (General disorders) | 20 | 20
hyperactivity (Nervous system disorders) | 10 | 7
impaired learning (Social circumstances) | 32 | 30
impulsivity (Social circumstances) | 12 | 21
insomnia (General disorders) | 27 | 28
libido changes (General disorders) | 6 | 8
nausea (Gastrointestinal disorders) | 11 | 15
numbness of fingers, toes, nose, ears, lips (Nervous system disorders) | 13 | 23
muscle stiffness or aching, muscle tenderness (Musculoskeletal and connective tissue disorders) | 38 | 40
palpitations (Cardiac disorders) | 8 | 5
skin rash, redness, or inflammation (Skin and subcutaneous tissue disorders) | 19 | 21
tachycardia (increased heart rate) (Cardiac disorders) | 3 | 6
urine color changes (Renal and urinary disorders) | 8 | 7
urine output, decreased (Renal and urinary disorders) | 7 | 7
unintentional weight loss (Metabolism and nutrition disorders) | 14 | 8
cough/congestion/bronchitis (Respiratory, thoracic and mediastinal disorders) | 12 | 11
diarrhea (Gastrointestinal disorders) | 10 | 8
falls with/without bruising (Injury, poisoning and procedural complications) | 10 | 6
feeling cold (Vascular disorders) | 0 | 6
fluid retention/swollen feet (General disorders) | 5 | 3
irritability (Nervous system disorders) | 4 | 8
night sweats (General disorders) | 0 | 5
pruritis (Skin and subcutaneous tissue disorders) | 5 | 2
Lost more than 7% of baseline body weight (Metabolism and nutrition disorders) | 10 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-25): https://cdn.clinicaltrials.gov/large-docs/01/NCT02346201/Prot_SAP_000.pdf